CLINICAL TRIAL: NCT06801795
Title: Evaluation of a 1726nm Laser for the Treatment of Hidradenitis Suppurativa (HS)
Brief Title: Aviclear for Hidradenitis Suppurativa (HS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ariel Eva Eber, Assistant Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240356
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- AviClear Group (Experimental): Participants will be in this group for up to 43 weeks.
  Interventions: Device: AviClear

INTERVENTIONS:
Device: AviClear — Participants will receive as many as 4 treatments, each treatment lasts approximately 10 minutes, with intervals of up to 5 weeks apart. The treatments will be conducted in person. Participants will be followed at approximately week 5 post-treatment completion (via phone) at 12 weeks and 24 weeks post treatment completion onsite.
  This is a 1726 nanometer laser treatment

SUMMARY:
The objective is to evaluate the safety and efficacy of the Cutera 1726 nm laser system (also referred to as AviClear) for the treatment of HS.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male.
2. Fitzpatrick Skin Types I-VI.
3. 18 to 60 years of age.
4. Has a clinical diagnosis of HS (stage 1-2 on the Hurley scale [Appendix 1] based on assessment by the investigator).
5. Presence of nodule(s) in the bilateral axillas, inguinal, infra-mammary, thighs, or buttocks within the past 4 weeks
6. Subject must be able to read, speak, and understand English or Spanish and sign the Informed Consent Form.
7. Willing and able to adhere to the treatment and follow-up schedule and pre/post-treatment care instructions.
8. No contraindication to laser therapy.
9. Willing to undergo biopsy at the beginning of study and end of study.
10. Willing to have photographs taken of the treatment area and agree to the use of photographs for presentation, educational or marketing purposes.
11. Agree to not undergo any other procedure(s) or add any new treatment modalities in the treatment area during the study.
12. Willing to use investigator approved skincare topicals and follow investigator approved skincare regimen for the duration of the study.

Exclusion Criteria:

1. Has clinically diagnosed HS of severity grade 3 based on assessment by the investigator.
2. Absence of nodule(s) in the bilateral axilla, inguinal, infra-mammary, thighs, or buttocks within the past 4 weeks.
3. Prior treatment to the target area during participation in a clinical trial of another device or drug within 1 month (30 days) prior to study participation.
4. Prior treatment to the target area within 3 months of study participation including chemical peel, dermabrasion, microneedling, radiofrequency treatment, laser or light-based procedures, cryodestruction or chemodestruction, intralesional steroids, photodynamic therapy, or acne surgery.
5. Prior injection of botulinum toxin in the target area within 3 months of study participation and for the duration of the study.
6. Systemic use of retinoid, such as isotretinoin, within 3 months of study participation.
7. Still healing from another treatment in the target area according to investigator's discretion.
8. History of malignant tumors in the target area.
9. Excessive hair that may preclude treatments, photos or accurate HS assessments in the target area (okay if shaved).
10. Pregnant and/or breastfeeding or planning to become pregnant during the study.
11. Suffering from diagnosed coagulation disorders or taking prescription anticoagulation medications.
12. History of diagnosed immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
13. History of diagnosed connective tissue disease, such as systemic lupus erythematosus or scleroderma.
14. Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
15. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the target area, unless treatment is conducted following a prophylactic regimen.
16. History of radiation to the target area, currently undergoing treatment for skin cancer in the target area or undergoing systemic chemotherapy for the treatment of cancer.
17. History of diagnosed pigmentary disorders (including vitiligo) in the target area.
18. Excessively tanned in the treatment area or unable/unlikely to refrain from tanning in the target area during the study.
19. History of keloids or hypertrophic scarring
20. Prisoners
21. As per the Investigator's discretion, any physical, mental or medical condition which might make it unsafe for the subject to participate in this study, might interfere with patient's participation in the full study protocol, or might interfere with the diagnosis or assessment of HS.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in HiSCR50 as measured by percentage of participants | Baseline, up to 24 weeks (after final treatment)
  Percentage of participants achieving Hidradenitis Suppurativa Clinical Response 50 (HiSCR50, where HiSCR50 is defined as at least a 50% reduction from baseline in abscess and inflammatory nodule (AN) count, with no increase from baseline in abscess or draining fistula count.

SECONDARY OUTCOMES:
Change in pain as measured by Visual Analogue Scale Pain Rating Scale | Baseline, up to 24 weeks (after final treatment)
  Score range from 0 to 10. Higher score indicates more pain.
Change in number of lesions | Baseline, up to 24 weeks (after final treatment)
  Number of lesions
Change in IHS 4 | Baseline, up to 24 weeks (after final treatment)
  The International Hidradenitis Suppurativa 4 (IHS 4) score is calculated as follows: number of nodules (multiplied by 1) + number of abscesses (multiplied by 2) + number of draining tunnels (multiplied by 4). A total score of 3 or less signifies mild, 4 to 10 signifies moderate, and 11 or higher signifies severe disease.
Change in number of Patient's stage category as measured by Hurley Stage | Baseline, up to 24 weeks (after final treatment)
  The unit of measure for this outcome is the change in number of patient's stage category. The different Hurley Stages are as follows:
  Patient's stage category I: Single of multiple abscess formation without sinus tracts and cicatrization Patient's stage category II: Recurrent single or multiple abscesses, widely separated, with limited sinus tracts and cicatrization Patient's stage category III: Diffuse or near-diffuse involvement of multiple interconnected tracts and abscesses across an entire area

CONTACTS AND LOCATIONS:
Overall Officials: Ariel E Eber, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No